CLINICAL TRIAL: NCT03882879
Title: Karate Intervention to Change Kinematic Outcomes in Parkinson's Disease. KICK OUT 2: A Phase Two, Randomized Trial of a Karate Intervention
Brief Title: Kick Out Parkinson's Disease 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 18012313-02
Record Dates: First submitted 2019-03-19; First posted 2019-03-20 (Actual); Results first posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2023-10

CONDITIONS: Parkinson Disease
Keywords: karate; exercise; martial arts; Parkinson's Disease; non-pharmacologic; randomized trial; camaraderie; depression; anxiety; quality of life
MeSH Terms: conditions — Parkinson Disease; Motor Activity; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This is a randomized, single-blinded, study of a novel intervention, namely, non-contact karate, for early to middle stage PD.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Participants in Arm 1 will begin participation in 6 months of karate classes immediately after the pre-intervention study visits.
  Interventions: Behavioral: Karate Classes; Behavioral: Pre-Intervention Study Visit; Behavioral: Bimonthly Online Survey; Behavioral: 6-month Study Visit; Behavioral: 12-month Study Visit
- Arm 2 (Experimental): Participants in Arm 2 will continue their usual exercise routine for six months followed by karate classes for six months
  Interventions: Behavioral: Karate Classes; Behavioral: Pre-Intervention Study Visit; Behavioral: Bimonthly Online Survey; Behavioral: 6-month Study Visit; Behavioral: 12-month Study Visit

INTERVENTIONS:
Behavioral: Karate Classes — Eligible subjects will engage in twice-weekly karate classes for 6 months, specifically designed for individuals with early to middle stage PD, focused on incorporating upper and lower limb movements in multiple directions, increasing awareness throughout the body, shifting body weight and rotation, relaxation of the muscles, improving reaction time, using complex repetitive actions to improve coordination, footwork training and centered weight shifts to help with fall prevention, and striking shields for self-defense and stress relief
Behavioral: Pre-Intervention Study Visit — At the pre-intervention study visit, the study logistics will be reviewed, informed consent process will occur, the subject will complete a battery of pre-intervention assessments focused on overall mobility, gait, balance, mood, cognition, and quality of life, and the subjects will be prompted to share their expectations of and goals for the karate classes.
Behavioral: Bimonthly Online Survey — All participants in both arms will receive a personalized email every two months directing them to indicate how frequently they have attended karate classes, how frequently they have engaged in exercise, how frequently they have fallen, whether their PD medication regimen has changed, and they will complete brief surveys about mood, camaraderie, and overall quality of life.
Behavioral: 6-month Study Visit — All participants in both arms will complete questionnaires and assessments of their PD symptoms, cognition, mood, camaraderie, and quality of life. Subjects will meet with a member of the study team to complete a series of physical and cognitive assessments. At this visit, subjects will review the initial expectations they shared at the pre-intervention visit and indicate if they thought their goals were achieved for the class.
Behavioral: 12-month Study Visit — At the 12-month study visit, the assessments from the baseline and 6-month study visit will be readministered, along with an assessment of the subject's global impression of change. Subjects will be prompted to share their thoughts on how the intervention impacted their overall wellbeing, balance, and mindfulness; whether the intervention achieved their expectations; and they will be asked to provide feedback for improvements.

SUMMARY:
The benefits of exercise for general health and well-being in older adults are well-established. Balance exercises such as tai chi and yoga, along with resistance training, can improve or maintain physical function in older adults and enhance muscle strength. Furthermore, aerobic activity is critical for maintaining and improving cardiovascular and functional health. Non-contact boxing has recently seen a surge in popularity among individuals with Parkinson's Disease (PD), with components of both aerobic and balance exercise. While participants anecdotally note improvements in stress and physical function, this has only been minimally studied. Therefore, we conducted a 10-week long pilot study of a structured karate exercise program. Among 15 participants, our pilot data highlights improvements in quality of life and high enthusiasm for the karate classes. Based on these promising results from the pilot, we are recruiting a larger, randomized group for the second phase of the karate intervention. The aim of this study is to test whether and to what degree a community-based karate class tailored for individuals with early- to middle-stage Parkinson's Disease (PD) 1) is feasible; 2) improves objective outcomes such as mobility and balance; 3) improves patient-reported outcomes compared with individuals given a standard exercise prescription for PD.

DETAILED DESCRIPTION:
For 6 months, eligible subjects will engage in twice-weekly karate classes, specifically designed for individuals with early to middle stage PD, focused on incorporating upper and lower limb movements in multiple directions, increasing awareness throughout the body, shifting body weight and rotation, relaxation of the muscles, improving reaction time, using complex repetitive actions to improve coordination, footwork training and centered weight shifts to help with fall prevention, and striking shields for self-defense and stress relief.

Due to both the capacity of the karate classes and the scientific approach to detecting changes in PD, subjects will be randomly assigned into either Arm 1: immediate participation in the karate class or Arm 2: participation in usual exercise for six months followed by karate classes for six months. For participants in Arm 1, following the first six months of classes, subjects may choose to continue their participation in karate and in the study, though this will require paying membership fees at the karate studio. For participants in Arm 2, following the first six months of usual exercise, participants will then begin 6 months of twice-weekly classes.

Before beginning the karate classes, each subject will attend a pre-intervention study visit during which subjects will complete assessments focused on overall mobility, gait, balance, mood, and quality of life. Subjects will receive a one-time, in-person training in best practices for exercise in PD. Also subjects will be prompted to share their expectations and goals for the karate classes.

All participants in both arms will receive a personalized email every two months directing them to indicate how frequently they attended karate classes or engaged in exercise, and they will complete assessments of mood and quality of life.

Following six months of classes for Arm 1, and six months of usual exercise for Arm 2, subjects will meet with the study team to complete assessments of mobility, gait, balance, mood, and quality of life. Arm 1 will participate in a focus group to review initial expectations and goals for the class.

The 12-month study visit will occur once Arm 1 and Arm 2 have completed the intervention. The assessments from the pre-intervention and 6-month study visit will be repeated. Subjects will participate in a focus group to share their thoughts on whether they would recommend the classes and how to improve the overall experience.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be those diagnosed with Parkinson's Disease by a treating healthcare provider; if the subject is seen at Rush University Medical Center, this will be verified via chart review. If the subject is seen elsewhere, he or she will be asked to have their a healthcare provider sign a form confirming the diagnosis of Parkinson's Disease and indicating that the subject can ambulate independently as of the most recent visit, to be sent back to the research coordinator for eligibility verification.
* English speaking
* Living within the Chicago area
* Subjects may be untreated for Parkinson's Disease, or may be taking any individual PD medication or combination thereof. Subjects may or may not have had Deep Brain Stimulation. Subjects may or may not be receiving physical or occupational therapy. Subjects will be encouraged to maintain their same medication regimen throughout the duration of the study, however if issues arise requiring medication changes, the subject will be prompted to indicate medication changes in the bimonthly online survey, and will not be disqualified from study participation.

Exclusion Criteria:

* Subjects requiring an assistive device (cane, walker, wheelchair) or the assistance of another person in order to ambulate.
* Subjects with active psychosis or exhibiting symptoms of a severe psychiatric disorder.
* Subjects unable to commit to attending, or to travel to, two classes weekly for 6 months.
* Subjects previously participating in a karate or other martial arts program, including boxing programs for PD, in the past 30 days.
* Subjects with atypical parkinsonism, including Progressive Supranuclear Palsy, Multiple System Atrophy, Dementia with Lewy Bodies, Corticobasal Syndrome, drug-induced parkinsonism, vascular parkinsonism, or atypical parkinsonism not otherwise specified, according to the referring healthcare provider.

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-03-03 (Actual); Primary Completion 2020-03-27 (Actual); Study Completion 2020-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jori Fleisher, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Baseline study visit and assessments completed after enrollment and prior to randomization.
Groups:
- Arm 1: Participants in Arm 1 will begin participation in 6 months of karate classes immediately after the pre-intervention study visits.
  Karate Classes: Twice-weekly karate classes for 6 months, specifically designed for individuals with early to middle stage PD.
  Pre-Intervention Study Visit: battery of pre-intervention assessments focused on overall mobility, gait, balance, mood, cognition, and quality of life, and the subjects will be prompted to share their expectations of and goals for the karate classes.
  Bimonthly Online Survey: how frequently they have attended karate classes, engaged in exercise, and fallen; and whether their PD medication regimen has changed. Brief surveys about mood, camaraderie, and overall quality of life.
  6-month Study Visit: Questionnaires and assessments of PD symptoms, cognition, mood, camaraderie, and quality of life; series of physical and cognitive assessments. Subjects will review the initial expectations they shared at the pre-intervention visit and indicate if they thought their goals were achieved for the class.
  12-month Study Visit: Assessments from the baseline and 6-month study visit will be readministered, plus subject's global impression of change.
- Arm 2: Participants in Arm 2 will continue their usual exercise routine for six months followed by karate classes for six months
  Karate Classes: Twice-weekly karate classes for 6 months, specifically designed for individuals with early to middle stage PD.
  Pre-Intervention Study Visit: battery of pre-intervention assessments focused on overall mobility, gait, balance, mood, cognition, and quality of life, and the subjects will be prompted to share their expectations of and goals for the karate classes.
  Bimonthly Online Survey: how frequently they have attended karate classes, engaged in exercise, and fallen; and whether their PD medication regimen has changed. Brief surveys about mood, camaraderie, and overall quality of life.
  6-month Study Visit: Questionnaires and assessments of PD symptoms, cognition, mood, camaraderie, and quality of life; series of physical and cognitive assessments. Subjects will review the initial expectations they shared at the pre-intervention visit and indicate if they thought their goals were achieved for the class.
  12-month Study Visit: Assessments from the baseline and 6-month study visit will be readministered, plus subject's global impression of change.
Period: Overall Study
Arm/Group | Arm 1 | Arm 2
Started | 27 | 25
6-month Visit | 19 | 20
Completed | 18 | 12
Not Completed | 9 | 13

BASELINE CHARACTERISTICS:
Population: Fifty two individuals enrolled; randomized 27 (Arm 1) to 25 (Arm 2)
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 27 | 25 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.56 (8.98) | 65.94 (9.82) | 65.74 (9.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 17 | 15 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 23 | 24 | 47
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 18 | 21 | 39
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 27 | 25 | 52
Prior experience in karate [Count of Participants; unit: Participants] | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Mobility as Measured by the Timed Up & Go (TUG)
Description: The Timed Up & Go (TUG) is a well-validated, brief measure of mobility. To complete this assessment, subjects sit in a standard arm chair and are instructed that when the team member says "Go", they should stand up from the chair, walk at their normal pace to a taped line, turn, walk back to their chair at a normal pace, and sit down again. The study team member will record the TUG results in seconds using a stopwatch. A lower TUG result indicates greater mobility. Scores at the pre- and post-intervention focus groups will be compared.
Time Frame: 12 months
Population: Participants evaluated at 12 month study visit.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 18 | 12
seconds
  Baseline | 9.66 (1.62) | 9.19 (1.56)
  12-month | 10.9 (1.67) | 10.03 (2.2)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; Test type: Superiority; p = 0.64, t-test, 2 sided

2. Secondary Outcome: Change in Overall Well-being as Measured by the Patient Global Impression of Change Scale (PGIC)
Description: The Patient Global Impression of Change Scale (PGIC) is a single-item rating scale that asks subjects to rate their overall response to the intervention using a 7-point rating scale, where 1 is "very much worse", 4 is "no change", and 7 is "very much improved". Percentages of subjects endorsing each of the 7 response options will be compared. This scale will be completed at the post-intervention focus group.
Time Frame: 12 months
Population: 17 participants in arm 1 and 12 in arm 2 completed PGIC scale; means compared at 12 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 17 | 12
score on a scale | 5.47 (1.18) | 5.75 (1.14)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; Test type: Superiority; p = 0.53, t-test, 2 sided

3. Other Pre Specified Outcome: Changes in Depression as Measured by the Hospital Anxiety and Depression Scale
Description: The Hospital Anxiety and Depression Scale is a brief, 14-item highly validated scale for measuring anxiety (7 items) and depression (7 items), with each item scored 0-3, and reverse scoring for negatively framed items. Scores for each subscale are totaled and categorized as normal (0-7 points), borderline abnormal (8-10 points), and abnormal (11-21) points. Scores at the pre-intervention, 6-month, and 12-month study visits will be compared.
Time Frame: 12 months
Population: 17 participants in arm 1 and 12 in arm 2 completed HADS at both baseline and 12 months. Difference within- and between-groups at 12 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 17 | 12
score on a scale
  Baseline | 4.53 (3.18) | 4.08 (3.23)
  12 months | 3.59 (2.62) | 2.92 (2.94)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; Test type: Superiority; p = 0.76, t-test, 2 sided — Between-group two-sided t-test

4. Other Pre Specified Outcome: Change in Quality of Life as Measured by the Parkinson's Disease Questionnaire- Short Form (PDQ-8)
Description: The Parkinson's Disease Questionnaire- Short Form (PDQ-8) is validated and shortened version of the PDQ-39, with 8 items each representing one domain of the PDQ-39, also with a summary index score standardized to a scale of 0-100, with higher scores signifying worse quality of life; this scale is recommended for use in PD by the Movement Disorder Society.
Time Frame: 12 months
Population: Participants completed the measure at baseline, 6, and 12 months. Analysis here includes within- and between-group differences at 12 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 18 | 12
score on a scale
  Baseline | 25.22 (16.73) | 29.25 (20.34)
  12-month | 20.67 (13.66) | 21 (17.58)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; Test type: Superiority; p = 0.49, t-test, 2 sided

5. Other Pre Specified Outcome: Change in Cognitive Domains as Measured by Montreal Cognitive Assessment
Description: A screening instrument designed to help health professionals detect mild cognitive dysfunction. Subjects will answer questions to measure different areas of cognition including attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. The total possible range is 0 (severely cognitively impaired) to 30 (perfect), where scores 26 and higher indicate normal cognition, and scores less than 26 indicate mild cognitive impairment or dementia.
Time Frame: 12 months
Population: 16 participants in arm 1 and 12 in arm 2 had MoCA data complete at both baseline and 12 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 16 | 12
score on a scale
  Baseline | 25.88 (2.66) | 26.67 (3.14)
  12 months | 25.88 (2.68) | 25.58 (3.15)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; Test type: Superiority; p = 0.20, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 1 year
Description: No difference from clinicaltrials.gov description
Arm/Group | Arm 1 | Arm 2
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/25
Serious Adverse Events (participants affected / at risk) | 2/27 | 1/25
Other Adverse Events (participants affected / at risk) | 0/27 | 1/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=27) | Arm 2 (N=25)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) — Urinary tract infection; deemed unrelated to study.
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Deemed unrelated to study
Surgery (General disorders) | 0 (0) | 1 (1) — Family member reported participant had surgery out of state, would not disclose underlying condition. Study team attempted to reach participant four more times without response
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=27) | Arm 2 (N=25)
Foot injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Stress injury to foot

LIMITATIONS AND CAVEATS:
12-month study visits were initially scheduled in the weeks immediately before and after COVID lockdowns, such that many participants were unable to complete the 12-month visits in-person and the primary outcome (Timed Up and Go) could not be assessed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-19): https://cdn.clinicaltrials.gov/large-docs/79/NCT03882879/Prot_SAP_000.pdf